CLINICAL TRIAL: NCT06733571
Title: An Observational Study on Validity of DULK Score as a Tool for Early Diagnosis of Anastomotic Leakage in the Immediate Post-Operative Period After Elective Primary Intestinal Anastomosis
Brief Title: Assessing the Validity of Dulk Score in Identifying Anastomotic Leak in Early Postoperative Period
Acronym: DULK
Status: Completed | Type: Observational
Sponsor: Sawai Mansingh Medical College (Other Government)
Responsible Party: Principal Investigator, DARSHAN KUMAR RATHOR, Resident Doctor, Department of General Surgery, Sawai Mansingh Medical College
Other Study IDs: SawaiMansinghMC; INSTITUTE (Other: SMS MC)
Record Dates: First submitted 2024-12-04; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Anastomosis, Leaking
Keywords: ANASTOTIC LEAK, DULK SCORE; DULK SCORE; LEAK

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing elective intestinal anastomosis procedures: The SMS Medical College Elective Intestinal Anastomosis Cohort is a prospective cohort study that includes patients undergoing elective intestinal anastomosis procedures at the Department of Surgery, SMS Medical College, Jaipur. This cohort consists of 86 patients who underwent various types of elective bowel reconnection surgeries, including jejuno-jejunal, ileo-ileal, ileo-colic, and colo-colic anastomoses, as well as stoma closures, between [study period]. The cohort includes both male and female patients aged 18 years and older who provided informed consent to participate.
  The primary aim of this cohort study is to assess the incidence and risk factors of anastomotic leaks (AL)-a serious postoperative complication that can significantly impact patient outcomes. Detailed monitoring of preoperative conditions, surgical factors, and postoperative outcomes, the study aims to identify key risk factors associated with AL, including patient comorbidities

SUMMARY:
Anastomotic leak is a commonly seen post-operative complication in patients who undergo bowel anastomosis. The outcome of which can range from conservative management to re-exteriorisation of bowel loop. This apart from financial distress can cause psychological impact on patient and his/her family. Understanding the risk factors identified, such as age, chronic diseases, anemia, and surgical variables, can aid healthcare providers in risk assessment, preoperative optimization, and postoperative monitoring to reduce the occurrence of anastomotic leaks.

By implementing strategies to address these risk factors, healthcare systems can improve patient outcomes, reduce complications, and enhance the quality of care provided to individuals undergoing surgical procedures, ultimately contributing to better public health outcomes and healthcare resource utilization.

DETAILED DESCRIPTION:
Study Population This study was conducted on a cohort of 86 patients who underwent elective open intestinal anastomosis at SMS Medical College, Jaipur. The patient population consisted of 48 males (59%) and 38 females (41%). The average age of the participants was 42.68 years, with a broad age range that allowed for the analysis of age-related risk factors in relation to anastomotic leaks (AL).

Risk Factors Considered for Anastomotic Leaks (AL)

Age and Gender:

The study explored the relationship between age and the incidence of anastomotic leaks, particularly focusing on age groups above 60 years. Gender-related patterns were also assessed.

Chronic Diseases:

Patients with chronic conditions such as diabetes mellitus, hypertension, and malignancy were included to assess their role in the development of anastomotic leaks.

Immunocompromised Status:

Patients with compromised immune systems, including those undergoing chemotherapy or immunosuppressive therapy, were considered in the study.

Chronic Steroid Use:

The impact of chronic steroid use on anastomotic leak rates was evaluated.

Anemia and Hypoalbuminemia:

The study assessed anemia (hemoglobin levels <10 g/dL) and hypoalbuminemia (serum albumin levels <3 g/dL) as potential risk factors for anastomotic leaks.

Leukocytosis:

Leukocytosis (elevated white blood cell count) was also examined as a risk factor.

Surgical Factors Considered

Surgical Technique:

The study evaluated whether the type of surgical technique (hand-sewn vs. stapled anastomosis) influenced the occurrence of anastomotic leaks.

Location of Anastomosis:

The effect of the location of the anastomosis (e.g., distal vs. proximal) on the risk of leaks was considered.

Duration of Surgery:

The study examined whether longer surgeries (lasting over 4 hours) were associated with a higher incidence of leaks.

Surgeon Experience:

The impact of surgeon experience on leak rates was considered, focusing on procedures performed by residents versus consultants.

DULK Score and Leak Detection The DULK score, a clinical scoring system, was used in the study to predict the likelihood of an anastomotic leak in the early postoperative period. Its role in identifying high-risk patients was an important aspect of the study.

ELIGIBILITY:
Inclusion Criteria:1. Patients who provided informed consent to participate in the study.

2. Patients aged 18 years or older. 3. Patients who underwent elective intestinal anastomosis in a planned operation (elective OT).

4. Patients with a single-site intestinal anastomosis.

-

Exclusion Criteria:1. Patients operated on in an emergency setting. 2. Patients who underwent anastomosis at multiple sites (e.g., multiple bowel resections, whipples operation).

3. Patients lost to follow-up during the post-operative period. 4. Patients who were unable or unwilling to provide informed consent. 5. Pregnant or breastfeeding women, as the study interventions may not be suitable during these periods.

6. Patients with significant cognitive impairments or psychiatric disorders that would limit their ability to understand the study protocol or provide informed consent.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study focused on patients undergoing elective intestinal anastomosis procedures at the Department of Surgery, SMS Medical College in Jaipur. These procedures included jejuno-jejunal, ileo-ileal anastomoses, ileo-colic and colo-colic anastomoses, as well as stoma closure. Prior to the surgeries, written informed consent was obtained from the patients. By specifically examining these elective procedures involving various types of anastomoses and stoma closure, the study aimed to investigate and analyse outcomes related to these surgical interventions within the clinical setting of the SMS Medical College in Jaipur.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-05-12 (Actual)

PRIMARY OUTCOMES:
ANASTOMOTIC LEAK | 12 DAYS
  The primary outcome measure is the incidence of anastomotic leaks (AL) in patients who undergo elective intestinal anastomosis at SMS Medical College, Jaipur. AL is defined as the failure of the bowel anastomosis to properly heal, leading to the leakage of intestinal contents into the peritoneal cavity, which may result in peritonitis or sepsis. The incidence is assessed in the postoperative period, primarily within the first 12 days following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Prabha OM, Study Chair — HOD DEPT OF GENERAL SURGERY
Locations (1):
- Sawai Man Singh Medical College, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: No
At this stage, the decision regarding whether to share individual participant data (IPD) with other researchers has not been finalized. We are currently evaluating the ethical, legal, and logistical considerations surrounding data sharing, including patient privacy, consent, and institutional guidelines. The primary goal is to ensure that any data shared respects participant confidentiality and complies with relevant regulations. If the decision is made to share the data, it will be made available through a secure platform, with proper oversight and approval from the relevant ethics committees. Further details will be provided once the final decision is made.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT06733571/Prot_SAP_000.pdf